CLINICAL TRIAL: NCT04362969
Title: Clinical Characteristics of Patients With SARS-CoV-2 (COVID-19) Infection in Guayaquil, Ecuador: COVID-EC Study
Brief Title: COVID-EC Study: Clinical Characteristics of Patients With COVID-19 in Guayaquil, Ecuador
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Universidad Catolica Santiago de Guayaquil (Other)
Responsible Party: Principal Investigator, Jorge Carriel M., Physician, Hospital San Carlos, Madrid
Other Study IDs: 001
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In December 2019, an outbreak of pneumonia of initially unknown cause was detected in Wuhan (Hubei, China), and it was quickly determined that it was caused by a new coronavirus, that is, the SARS-CoV- 2 virus, causing the disease called COVID-19. Since then, the outbreak has spread to 5 continents, affecting 185 countries or regions, with more than 2,500,000 confirmed cases as of April 21, 2020. Ecuador, the 9th country according to territorial extension, and the 7th according to the number of inhabitants in South America, is the 4th country with the highest number of cases in that region of the world, only behind Brazil, Peru and Chile. According to data from the Ministry of Public Health (MSP) of Ecuador, as of April 20, 2020, the National Institute for Public Health Research (INSPI) has registered 33,279 samples, of which 10,128 are positive for SARS-CoV-2. By far, the province of Guayas where Guayaquil is located, the main city in terms of number of inhabitants of the country, is the region with the highest number of affected, with 6921 confirmed cases and 6274 with suspicion.

Given the importance of this infection, the severity in some cases, its rapid distribution, and the differences in the Ecuadorian population with respect to the other countries where infected patients have been reported, the investigators consider that an updated analysis of cases, taking as a reference, patients seen in various hospitals of the city of Guayaquil can help identify the clinical characteristics and severity of the disease.

DETAILED DESCRIPTION:
Design: Retrospective cohort study that will review the data of patients seen in participating centers with a confirmed or probable diagnosis of COVID-19 between March and April 2020. Those patients who test positive for nasopharyngeal exudate for SARS-CoV-2 will be considered a confirmed case using the real-time reverse transcriptase polymerase chain reaction (RT-PCR) technique. A patient with a severe acute respiratory infection (with fever and who needs to be hospitalized), and without another etiology that fully explains the clinical manifestations, and who has traveled to or resided in China in the 14 days prior to the onset of symptoms, or a patient with any acute respiratory illness and in whom at least one of the following conditions is met in the last 14 days prior to the onset of symptoms: having contact with a confirmed or probable case of infection with the COVID-19 virus, or having worked or been in a health care facility where patients with confirmed or probable infection with the COVID-19 virus were being treated, according to WHO criteria. Cases with nasopharyngeal exudate for SARS-CoV-2 negative are excluded from the study.

Ambit: Emergency, hospitalization and intensive care services at participating centers.

Subjects to study: Patients older than 18 years with a confirmed or suspected diagnosis of COVID-19 that required admission at participating centers.

Study variables:

* Demographic variables: Age, Sex, Personal history (hypertension, diabetes, previous cardiovascular disease, previous chronic lung disease, active smoking, obesity, etc.).
* Clinical variables: previous contact with a confirmed or suspected COVID-19 patient, days of onset of symptoms until the first consultation, symptoms (fever, asthenia / deterioration of general condition, cough, dyspnea, anosmia, ageusia, diarrhea, nausea, headache), signs present in the first recorded physical examination (blood pressure, saturation, temperature, heart rate, respiratory rate, auscultation, edema, weight and height).
* Laboratory variables: blood count, C-reactive protein (PCR), procalcitonin (PCT), lactate dehydrogenase (LDH), D-dimer, Ferritin, AST, ALT, GGT, Alkaline phosphatase, coagulation times, creatinine, urea, sodium, potassium . Arterial blood gas when available.
* Radiological variables: findings on plain radiography and chest computed tomography (CT).
* Microbiological variables: nasopharyngeal exudate for SARS-CoV-2, sputum culture, bronchoalveolar lavage, blood cultures, urine culture.
* Prognostic variables: need for hospitalization, length of hospital stay, need for admission to the Intensive Surveillance Unit (LVU), length of stay at LVU, need for invasive or non-invasive mechanical ventilation (MV), development of respiratory distress syndrome (ARDS), pneumonia, severity of pneumonia (CURB-65), sepsis (qSOFA), renal failure, electrolytic disturbances, stroke, ischemic heart disease, pulmonary embolism (PE) or deep vein thrombosis (DVT) and death.
* Therapeutic variables: treatment administered (Hydroxychloroquine, Chloroquine, Azithromycin, Lopinavir / Ritonavir, Oseltamivir, Tocilizumab, Corticosteroids, Ivermectin, Nitaxozanide, Enoxaparin or other low molecular weight heparin), dose administered, drug combination, time of administration, (counting the days from the onset of symptoms), registered adverse effects.

Definitions: Fever is defined as axillary temperature greater than 37.5ºC. Lymphopenia is defined as the presence of <1500 cells / mm3. Thrombocytopenia is defined as the presence of <150,000 platelets / mm3. ARDS will be defined according to the Berlin criteria, CID according to the ISTH criteria, Pneumonia will be defined according to SEPAR criteria and its severity will be based on the CURB-65 scale. The rest of the variables that require a definition will be defined according to standard clinical practice.

Statistic analysis: The data will be collected in a Microsoft Excel database, and will be exported to the SPSS statistical package for mathematical analysis. The mean and standard deviation (SD) will be used as measures of centralization and dispersion, respectively, in the case of quantitative variables with normal distribution. In case of variables that do not present normal distribution, the median and the interquartile range (RIQ) will be used. The study of the normality of the distributions will be carried out using the Kolmogorov-Smirnov test. Qualitative variables will be expressed as percentages.

-Inferential: The independent means will be compared using the Student's t test for variables that follow a normal distribution, otherwise the Mann-Whitney U test will be used. The Wilcoxon test will be used for paired data. The association between qualitative variables will be evaluated by means of the Chi square test (χ2) (or Fisher's test, if applicable). In the hypothesis test it will require an error α less than 0.05 to reject the null hypothesis.

Ethical aspects: In the process and development of the present study, patients will not be contacted and only the information collected in the medical records will be accessed. These medical records will be used solely and exclusively for the purposes of the study.

The study presented here will follow the standards of Good Clinical Practice, the principles of the Declaration of Helsinki (Seoul 2013), and the Oviedo Convention (1997). No identifying or clinical data of the patients will be provided and the investigators will work on an anonymized and password protected file that does not allow traceability of the people included in the registry. Likewise, the handling of data will be carried out in accordance with the provisions of the Law on data protection and the Law on the rights and protection of the patient.

Informed consent: The investigators will request exemption from informed consent as it is considered disproportionate measures to call or make appointments for each of the patients or their families, taking into account that this is a retrospective study based on the review of medical records. The database will be anonymized in compliance with current legal regulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older who required hospitalization.
* Confirmed diagnosis of COVID-19 by positive nasopharyngeal exudate for SARS-CoV-2.
* Probable diagnosis of COVID-19, according to WHO criteria.

Exclusion Criteria:

- Patients with negative nasopharyngeal exudate for SARS-CoV-2.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult population hospitalized by COVID-19 in public and private hospitals in the city of Guayaquil, Ecuador.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of patients with COVID-19 | 4 weeks
  To know the clinical characteristics of patients with COVID-19 treated in hospitals in Guayaquil, Ecuador.

SECONDARY OUTCOMES:
Prognosis of patients, in terms of need for admission to intensive care, use of mechanical ventilation or death | 4 weeks
  Establish the prognosis of patients, in terms of need for admission to intensive care, use of mechanical ventilation or death.
Clinical characteristics of the patients with the worst prognosis | 4 weeks
  To determine the clinical characteristics of the patients with the worst prognosis.
Relationship between the different treatments and the prognosis | 4 weeks
  Relate, at least retrospectively, the relationship that may exist between the different treatments and the prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: JORGE CARRIEL, Principal Investigator — Hospital Clínico San Carlos, Madrid
Locations (1):
- GastroMuñoz, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Background] Boletín No 053 con fecha 20/04/2020 del Ministerio de Salud Pública sobre COVID-2019 Ecuador [Internet]. 2020 [cited 2020 Apr 21]. Available from: https://www.salud.gob.ec/wp-content/uploads/2020/04/Boletin-053-AM_Nacional.pdf
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Ki M; Task Force for 2019-nCoV. Epidemiologic characteristics of early cases with 2019 novel coronavirus (2019-nCoV) disease in Korea. Epidemiol Health. 2020;42:e2020007. doi: 10.4178/epih.e2020007. Epub 2020 Feb 9. PMID 32035431
- [Background] Wang Y, Lu X, Li Y, Chen H, Chen T, Su N, Huang F, Zhou J, Zhang B, Yan F, Wang J. Clinical Course and Outcomes of 344 Intensive Care Patients with COVID-19. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1430-1434. doi: 10.1164/rccm.202003-0736LE. No abstract available. PMID 32267160
- [Background] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] OMS. Protocolo de investigación de los primeros casos y sus contactos directos (FFX) de la enfermedad por Coronavirus 2019 (COVID-19). 2020;2:1-83.
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Toh CH, Hoots WK; SSC on Disseminated Intravascular Coagulation of the ISTH. The scoring system of the Scientific and Standardisation Committee on Disseminated Intravascular Coagulation of the International Society on Thrombosis and Haemostasis: a 5-year overview. J Thromb Haemost. 2007 Mar;5(3):604-6. doi: 10.1111/j.1538-7836.2007.02313.x. Epub 2006 Nov 10. No abstract available. PMID 17096704
- [Background] Menendez R, Torres A, Aspa J, Capelastegui A, Prat C, Rodriguez de Castro F; Sociedad Espanola de Neumologia y Cirugia Toracica. [Community acquired pneumonia. New guidelines of the Spanish Society of Chest Diseases and Thoracic Surgery (SEPAR)]. Arch Bronconeumol. 2010 Oct;46(10):543-58. doi: 10.1016/j.arbres.2010.06.014. Epub 2010 Sep 15. No abstract available. Spanish. PMID 20832928
- [Background] Shah BA, Ahmed W, Dhobi GN, Shah NN, Khursheed SQ, Haq I. Validity of pneumonia severity index and CURB-65 severity scoring systems in community acquired pneumonia in an Indian setting. Indian J Chest Dis Allied Sci. 2010 Jan-Mar;52(1):9-17. PMID 20364609